CLINICAL TRIAL: NCT03231787
Title: Randomized Parallel Multicenter Trial in Antiaggregated Patients With Proximal Femur Fracture Evaluating a Strategy to Shorten Time Until Surgery (AFFEcT Study)
Brief Title: Clinical Trial in Antiaggregated Patients With Proximal Femur Fracture Evaluating a Strategy to Shorten Time Until Surgery
Acronym: AFFEcT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Carlos III Health Institute (Other Government); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIBSP-PLA-2016-86
Record Dates: First submitted 2017-07-19; First posted 2017-07-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In this group the platelet aggregability will be evaluated and if it is normal, the surgery will be performed within 24-48 hours.
  If it is not normal, the evaluation of platelet aggregability will be repeated daily until the third day or until it is normalized if it is earlier.
  If at the third day is not normalized, it will proceed as with the control group, which will take into account the safety time of the drug.
  Interventions: Diagnostic Test: Platelet function assay
- Control group (No Intervention): The control group will wait for the safety time of the drug according to the usual practice of the center.

INTERVENTIONS:
Diagnostic Test: Platelet function assay — Plateletworks is an in vitro diagnostic screening assay for the determination of % platelet aggregation or % platelet inhibition.
  It will be used to measure platelet function after withdrawal of the antiplatelet agent.
  If there are more than 80,000 functional platelets, the patient will be operated on within the next 24 hours.
  Other Names: Plateletworks®
  Arms: Experimental group

SUMMARY:
National, randomized, open, parallel, multicenter clinical trial of two comparison groups that will evaluate the feasibility of a strategy based on a diagnostic test to shorten the surgery time in antiaggregated patients with proximal femur fracture.

The experimental group will undergo surgery as soon as platelet aggregability, according to the PLATELETWORKS® method is correct within 24-48 hours.

The control group will undergo surgery according to the usual practice of the center taking into account the safety time of the antiplatelet agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients of both sexes
* Patients with a proximal femoral fracture requiring surgery
* Patients receiving antiplatelet agents at the time of admission to the emergency room: AAS> 100 mg / d (Aspirin®), Trifusal> 300 mg / d (Digren®; Edigen®), clopidogrel (Plavix®), prasugrel ®), ticagrelor (Brilique ®) and ticlopidine (Tiklid ®).
* Patients who give their signed consent

Exclusion Criteria:

* Multiple fractures
* Pathological fractures
* Patients receiving vitamin K antagonist oral anticoagulants (warfarin and acenocoumarol) or new oral anticoagulants (apixaban, rivaroxaban and dabigatran) or who have acquired congenital or acquired coagulopathy
* Patients with AAS ≤100mg, trifusal ≤300mg
* Patients who do not give their informed consent or their legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Time from emergency admission to surgery | Up to 120 hours
  Time from emergency admission to surgery will be measured in hours

SECONDARY OUTCOMES:
Bleeding | Through hospitalization, an average of 5 days
  Total blood loss calculated by Nadler's formula from date of surgery until date of discharge
Need for blood transfusion | Through hospitalization, an average of 5 days
  Need for blood transfusion during hospitalization and transfused units
Preoperative hemoglobin | 12 hours before surgery
  Measurement of preoperative hemoglobin during 12 h before surgery
Postoperative hemoglobin | From 12 hours after surgery until date of discharge, an average of 5 days
  Measurement of postoperative hemoglobin until discharge
Surgical wound complications | 1 week and 30 days after surgery
  It includes:
  * Wound infection
  * Wound dehiscence
  * Reoperation due to wound complications
  * Postoperative pain
  * Safety: including the incidence of deep venous thrombosis during admission
Medical complications | 1 week and 30 days after surgery
  Myocardial infarction, stroke, pulmonary embolism, pneumonia / respiratory infections, urinary tract infections, sepsis, new onset pressure ulcers, acute renal failure, heart failure, delirium.
Platelet Functionality | From date of admission until the day before surgery, an average of 2 days
  Measurement of platelet functionality with plateletworks
Quality of life | Preoperative, 5 days after surgery, and 1, 6 and 12 months after surgery
  Quality of life measured by EQ-5D-5L questionnaire
Time to admission to patient movilization | From date of admission until the date of first movilization, an average of 3 days
  Time to admission to patient movilization measured in days
Mortality | 1 year
  All causes mortality
Cost effectiveness ratio | 1 year
  Cost effectiveness ratio (Δ cost / Δ effectiveness)

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Martinez Zapata, MD, PhD, Principal Investigator — Institut de Recerca Hospital de la Santa Creu i Sant Pau - IIB Sant Pau
Locations (3):
- Spain (3):
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided